CLINICAL TRIAL: NCT01703416
Title: CorRELation Between PatIent PErception of the Ability to Perform Morning Activities and Findings on Clinical Examination in COPD Patients Receiving Inhaled Combined Therapy (Corticosteroid/Long Acting ß2-agonist) - RELIEF Study
Brief Title: Correlation Between Patient Perception and Findings on Clinical Examination in Chronic Obstructive Pulmonary Disease (COPD) Patients
Acronym: RELIEF
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RBG-ATC-2012/1
Record Dates: First submitted 2012-10-03; First posted 2012-10-10 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; GOLD group C and D; CDLM questionnaire; visual scale - physician evaluation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
This is a multi-center, prospective, non-interventional study that aims to evaluate in daily clinical practice the possible correlation between patient perception of the ability to perform morning activities and the physician's assessment during a regular physical exam in patients with Chronic Obstructive Pulmonary Disease (COPD), group C and D.

DETAILED DESCRIPTION:
CorRELation between PatIent PErception of the Ability to Perform Morning Activities and Findings on Clinical Examination in COPD Patients receiving inhaled combined therapy (corticosteroid/long acting ß2-agonist) - RELIEF Study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD), group C and D according to GOLD Guidelines, 2011
* Receive inhaled combined therapy for COPD (inhaled corticosteroid / long acting ß2-agonist); this treatment should have been initiated for at least one month before entering the study
* Current or past smokers, of at least 10 pack years

Exclusion Criteria:

* History of exacerbation of COPD symptoms within the last month before visit 1, inclusive.
* History of asthma or allergic rhinitis.
* History of lung carcinoma or any other respiratory condition that may limit the airflow circulation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Obstructive Pulmonary Disease (COPD) patients group C and D
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in CDLM (Capacity of Daily Living during the Morning) questionnaire. | Baseline and 3 months
Change from baseline of patient's general health status upon physical evaluation - visual scale | Baseline and 3 months

SECONDARY OUTCOMES:
Age (years), gender (male/female), weight (kg), height (cm), place of origin (urban/rural) | Day 0 (visit 1)
  Descriptive statistics will be calculated for this outcome measure
Number of daily walking steps (by using pedometers) | up to 3 months
Patient adherence to treatment (by using visual 5 point scale) | up to 3 months
Number of unscheduled visit (exacerbations, emergency visits) | up to 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- Bulgaria (2):
  - Sofia
  - Varna